CLINICAL TRIAL: NCT03635671
Title: Diabetic Retinopathy and Subclinical Signs of Disease Transition
Acronym: DIRECTION
Status: Terminated | Type: Observational
Why Stopped: Unexpected poor enrollment
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, David Maberley, MD, FRCSC, University of British Columbia
Other Study IDs: DIRECTION
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Retinopathy
Keywords: Imaging; Diabetes; OCTA
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensified blood glucose control: Patients with diabetes mellitus type 2 and poor blood sugar control that are introduced to insulin or GLP-1 therapy
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography
- Nephropathy: Patients that are introduced to hemodialysis or renal transplantation secondary to renal failure
  Interventions: Diagnostic Test: Optical Coherence Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography Angiography — Retinal scans will be acquired at each follow up visit
  Other Names: Optical Coherence Tomography

SUMMARY:
The prevalence of diabetes mellitus (DM) is increasing worldwide. Diabetic retinopathy is the most prevalent complication of DM and a leading cause of visual impairment. Some factors are known to temporarily aggravate or improve diabetic retinopathy, but underlying pathophysiologic factors are still unknown. High-resolution imaging techniques of the retina and its supplying vascular networks now allow novel insight to subtle changes that cannot be appreciated in standard fundus examination. In detail, the investigators image study patients with optical coherence tomography (OCT) - technology, that provides morphological information of retinal structure and the supplying vessels in a non-invasive way. Retinal layer thickness as well as capillary density will be quantified and followed in patients that are in a critical period of disease transition to better understand the process of diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2
* Age 18-90

Exclusion Criteria:

* Media opacities like cataract or vitreous hemorrhage
* Active intraocular inflammation (grade trace or above) in either eye like infectious conjunctivitis, keratitis, scleritis, endophthalmitis as well as idiopathic or autoimmune-associated uveitis in either eye
* Structural damage to the center of macula in the study eye
* Atrophy of retinal pigment epithelium, subretinal fibrosis, laser scar within foveal avascular zone (FAZ) or organized hard exudate plaques
* Ocular disorders in the study eye including retinal vascular occlusion, retinal detachment, macular hole, choroidal neovascularization, macula dystrophies
* Intraocular surgery (including cataract surgery, YAG laser capsulotomy) in the study eye within 3 months preceding Day 0, or history of corneal transplantation in the study eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with anti-glaucoma medication)or history of glaucoma filtration surgery
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes type 1 or 2 that enter a critical period of possible disease transition will be recruited in a tertiary referral center.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Perfusion density | 6 months
  Mean change of perfusion density of the macula evaluated within the 9 ETDRS subfields for the superior and inferior vascular plexus separately.

SECONDARY OUTCOMES:
Perfusion density | 12 months
  Mean change of perfusion density of the macula evaluated within the 9 ETDRS subfields for the superior and inferior vascular plexus separately.
Retinal layer thickness | 6 and 12 months
  Mean change in retinal layer thickness of all retinal layers separately

CONTACTS AND LOCATIONS:
Overall Officials: David Maberley, MD, Principal Investigator — Head of the Department of Ophthalmology and Visual Science, UBC
Locations (1):
- Eye Care Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No